CLINICAL TRIAL: NCT05252169
Title: Effects of Proprioceptive Training on Balance and Motor Function in Children With Spastic Hemiplegic Cerebral Palsy
Brief Title: Proprioceptive Training,Balance,Motor Function,Spastic Cerebral Palsy Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/1079/2021
Record Dates: First submitted 2022-02-12; First posted 2022-02-23 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-02

CONDITIONS: Hemiplegic Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive Training (Experimental): Proprioceptive training will include : Stair climbing up and down,Standing with feet side by side and up and down,one leg standing,Walking heel to toes,Rising from a standard chair.
  Swiss ball activity will be performed passively by the physical therapist in which child will sit on the ball and ball will be rolled from side to side,Extension rotation and flexion rotation will be performed to facilitate trunk rotation that will be performed with stabilized pelvis and hip.
  Routine physical therapy will include passive stretching ,strength training and weight bearing exercises. total session will be of 60 minutes.
  Interventions: Other: Proprioceptive training; Other: Routine Physical therapy
- Routine Physical Therapy (Placebo Comparator): Group A will be given routine physical therapy which will be of 60 minutes each session. The routine physical therapy will include
  * Passive stretching exercises
  * Weight bearing exercises
  * Functional strength training Duration of the treatment will be 3 days a week for 12 weeks i.e., 36 sessions. Each session will be of 60 minutes.
  Interventions: Other: Routine Physical therapy

INTERVENTIONS:
Other: Proprioceptive training — Proprioceptive Training will include some active exercises such as stair climbing up and down,one leg standing,Walking heel to toes,rising from a standard chair.
  And swiss ball training will be applied passively by therapist in which child will sit on the ball and ball will be rolled from side to side,Extension rotation and flexion rotation will be performed to facilitate trunk rotation,Trunk rotation will be performed with stabilized pelvis and hip.
  Other Names: Routine physical therapy
  Arms: Proprioceptive Training
Other: Routine Physical therapy — Group A will be given routine physical therapy which will be of 60 minutes each session. The routine physical therapy will include
  * Passive stretching exercises
  * Weight bearing exercises
  * Functional strength training Duration of the treatment will be 3 days a week for 12 weeks i.e., 36 sessions. Each session will be of 60 minutes.

SUMMARY:
Study Design: Randomized Controlled Trial Settings: Study will be conducted at Mobility quest clinic, Lahore Sample size:37 in each group Control group receive : Routine physical therapy Experimental group receive : Routine physical therapy+proprioceptive training

DETAILED DESCRIPTION:
Control group : Group A will be control group which will be of 60 minutes each session. The routine physical therapy will include

* Passive stretching exercises
* Weight bearing exercises
* Functional strength training Duration of the treatment will be 3 days a week for 12 weeks i.e., 36 sessions. Each session will be of 60 minutes.

Experimental group : Routine physical therapy+proprioceptive training. Group B will be given proprioceptive training. Duration of the treatment will be 3 days a week for 12 weeks i.e., 36 sessions. Each session will be of 60 minutes each session.

The Proprioceptive training included the following exercises.

* Stair climbing up and down (a regular 3 steps staircase).
* Standing with feet approximately shoulder-width apart and arms extended out slightly forward lower than the shoulder, then lifting both heel off the floor and to hold the position for 10 seconds, followed by climbing regular steps staircase. This procedure will be performed with eyes closed also.
* Standing with feet side by side & holding the arms in same position as described above, one foot is placed on the inside of the opposing ankle and to hold the position for 10 seconds. Followed by climbing regular steps staircase. This procedure will be performed will be eyes closed also.
* To perform one leg standing with one foot raised to the back and to maintain the position for minimum 3 seconds. This procedure will be performed with eyes closed also.
* Same exercise as above performed but with one foot raised to the front. This procedure will be then performed with eyes closed.
* Walking heel to toes.
* Rising from a standard chair (4 times) without arm support. For proprioception Swiss ball will be use as a modality and it will be performed passively by the physical therapist.For this physical therapist will be on the front of the subject different activities will be performed in different positions.
* For posture control development child will sit on the ball and ball will be rolled from side to side.
* Extension rotation and flexion rotation will be performed to facilitate trunk rotation.
* Trunk rotation will be performed with stabilized pelvis and hip. Reaching activities will be done in different directions that will allow the child to work on trunk and lateral weight shifting.
* Position the child supine on the ball with the feet to the floor. Hold through the lower abdominals to stabilize them on to the ball. Now facilitate through one arm and bring the child diagonally up to stance.

ELIGIBILITY:
Inclusion Criteria:

* • Children with spastic hemiplegic cerebral palsy ranging from 8 to 14 years. 19

  * Both genders.
  * Gross motor function level II.
  * Children who can follow commands.
  * Pre-diagnosed cerebral palsy subjects of cerebral palsy confirmed by an expert pediatrician.

Exclusion Criteria:

* • The children with cerebral palsy having co-morbid conditions and contractures that can interfere with recovery will be excluded.

  * The children having severe mental retardation because of difficulty in understanding commands.
  * Any red flag signs (tumor, fracture, metabolic diseases, prolong history of steroidal use.
  * Patients having ventriculoperitonel shunt.
  * Patients unable to travel frequently or as per call from rehab center.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2021-12-23 (Actual); Primary Completion 2022-08-16 (Estimated); Study Completion 2022-08-26 (Estimated)

PRIMARY OUTCOMES:
Balance | 12 weeks
  balance will be measured by pediatric balance scale.The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points.
Motor Function | 12 weeks
  Motor function will be measured by Gross Motor Function Measure 88 scale.It includes scoring key in which 0 means does not initiate and 3 means completely performs the exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Kinza Amin, MSPTN*, Principal Investigator — Univerity of Lahore
Locations (1):
- Mobility Quest Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown KE, Neva JL, Ledwell NM, Boyd LA. Use of transcranial magnetic stimulation in the treatment of selected movement disorders. Degener Neurol Neuromuscul Dis. 2014 Dec 4;4:133-151. doi: 10.2147/DNND.S70079. eCollection 2014. PMID 32669907
- [Background] Newbury DF, Simpson NH, Thompson PA, Bishop DVM. Stage 2 Registered Report: Variation in neurodevelopmental outcomes in children with sex chromosome trisomies: testing the double hit hypothesis. Wellcome Open Res. 2021 Jun 1;3:85. doi: 10.12688/wellcomeopenres.14677.4. eCollection 2018. PMID 30271887
- [Background] Uwizeye D, Karimi F, Thiong'o C, Syonguvi J, Ochieng V, Kiroro F, Gateri A, Khisa AM, Wao H. Factors associated with research productivity in higher education institutions in Africa: a systematic review. AAS Open Res. 2022 Jan 28;4:26. doi: 10.12688/aasopenres.13211.2. eCollection 2021. PMID 34368619
- [Background] Ozyurek T, Demiryurek EO. Comparison of the Effectiveness of Different Techniques for Supportive Removal of Root Canal Filling Material. Eur Endod J. 2016 Dec 26;1(1):1-6. doi: 10.5152/eej.2016.16002. eCollection 2016. PMID 32566900